CLINICAL TRIAL: NCT02282865
Title: The Relationship Between the Surgery-related Anxiety and HRV: Prediction for Aggressive Emergence Behavior
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0599
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Closed Reduction Surgery for Nasal Bone Fracture
Keywords: Emergence agitation, Heart rate variability (HRV)
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Visual analogue scale (VAS) >5: The degree of surgery-related anxiety assessment using VAS
- Visual analogue scale (VAS) ≤5: The degree of surgery-related anxiety assessment using VAS

SUMMARY:
Heart rate variability (HRV) is known to reflect the balance of autonomic nervous system. Anxiousness, which tend to result from the deficient action of parasympathetic nervous system, likely to show low HRV. This study is to investigate the relationship between the surgery-related anxiety and the HRV which is known to reflect the balance of autonomic nervous system. Furthermore, this study also focuses on HRV's role as a predictor for aggressive emergence behavior, which might also be considered as partially related to imbalance of autonomic nervous system.

ELIGIBILITY:
Inclusion Criteria:

1. 20-60 years old male, ASA 1-2
2. scheduled for elective closed reduction for nasal bone fracture

Exclusion Criteria:

1. Patients having hearing difficulties, Foreigner, taking any CNS related medication, history of any adverse drug reaction, Glasgow coma scale < 15
2. patients with severe cardiopulmonary dysfunction
3. patients taking any neurologic medication (anti-depressant, anti-convulsant, etc)
4. patients taking any cardiovascular medication
5. patients taking medications affecting the autonomic nervous system (a-blocker, b-blocker, etc)
6. patients refusal

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20-60 years old male, ASA 1-2, scheduled for elective closed reduction for nasal bone fracture.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2014-09-11 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
High frequency (HF) of Heart Rate Variability (HRV) | from immediately after tracheal intubation to 5 min after tracheal intubation
  High frequency (HF) component of HRV, which represents the parasympathetic activity

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea